CLINICAL TRIAL: NCT04646616
Title: CRISOL: Building Community Resilience and Integrating Efforts to Understand and Address Syndemic Health Conditions Afflicting Young LatinoImmigrants
Brief Title: CRISOL Contigo: a Multi-level Intervention to Reduce the Disproportionate Toll of COVID-19 Among Latino Communities in Philadelphia.
Acronym: CRISOL Contigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Ana Martinez Donate, Professor of Community Health and Prevention, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3R21MD012352-02S1 (NIH)
Record Dates: First submitted 2020-11-25; First posted 2020-11-30 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Covid19; Mental Health Issue; Violence
Keywords: Latino health; Immigrant health; Syndemic
MeSH Terms: conditions — COVID-19 | interventions — Genes, pol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community popular opinion leader (POL) (Experimental): After successful completion of the new COVID-19 training module, POLs will reach out to members of their social networks to model and diffuse social norms to reduce the risk of COVID-19 infection and transmission, screen for symptoms and counsel regarding COVID-19, SAVAME syndemic factors, and refer at-risk or affected individuals to appropriate community services (e.g. free COVID-19 testing and treatment, mental health services, substance use services, violence prevention, support groups, etc.). As in other POL based interventions and pragmatic trials, POLs be asked to follow up with their community contacts to monitor their situation and provide additional support, but there will be flexibility with the frequency and number of follow up contacts depending on their needs identified and the preferences of the community contact. POLs will be continually supported by the research team via face-to-face biweekly booster sessions (if COVID-19 situation requires it) or by zoom.
  Interventions: Other: Community popular opinion leader (POL) based intervention

INTERVENTIONS:
Other: Community popular opinion leader (POL) based intervention — A community popular opinion leader (POL) based intervention to promote measures to reduce COVID-19 risk, transmission, access to testing and treatment, reduction of the impact of COVID-19, and addressing the Substance Abuse, Violence, HIV/AIDS, and MEntal health (SAVAME) syndemic in the community. POLs will interact within their networks counseling regarding COVID-19 and SAVAME factors. The POLs will refer individuals to appropriate community services. POLs will record basic sociodemographic characteristics of all community contacts, the issue addressed, and their response to it. The first 300 community contacts will be invited to complete a baseline and 3-month follow up surveys (via internet or phone). The content of the surveys includes: 1) COVID-19 related questions (knowledge, impact, symptoms, risk factors, access to testing and care, acceptability contact tracing, vaccine) 2) Biological risk factors, 3) Social determinants of health, 4) SAVAME outcomes and access to services.

SUMMARY:
Latinos have been one of the racial/ethnic groups most impacted by the COVID-19 pandemic, and evidence of effective strategies to curb the pandemic, reduce disparities, and mitigate its impact is lacking and very urgent.

The goal of this competitive revision is to expand an ongoing academic-community partnership to adapt, implement, and evaluate a multi-level intervention to mitigate the multi-dimensional toll of COVID19 among Latino immigrant communities in Philadelphia.

DETAILED DESCRIPTION:
This goal of this competitive revision is to expand our original project to adapt, implement and evaluate a multi-level intervention to mitigate the multi-dimensional toll of COVID19 among Latino immigrant communities in Philadelphia. Evidence of effective strategies to curb the pandemic, reduce disparities and mitigate its impact is lacking and very urgent. In the US, Latino immigrants are one of the groups hardest hit by this pandemic, with recent steep increases in COVID-19 deaths among this group corroborating their continued increased risk of infection and increased susceptibility. Latino immigrants have long exhibited disparities in diabetes, obesity and hypertension, factors known to increase COVID-19 related severity, and also in Substance Abuse, Violence exposure, HIV/AIDS, and MEntal health (SAVAME) syndemic. These syndemic conditions have been worsened in the context of COVID-19. Latino immigrants represent a hard-to-reach and marginalized population, with extremely limited access to adequate health care and safety nets. This group faces many structural barriers, and social vulnerabilities, that hinder their capacity to access COVID-19 testing and treatment services and to adhere to public health interventions and measures to decrease the spread of COVID-19. Latinos often rely on a thin and fragmented network of health and social services organizations. Intervention to mitigate the impact of COVID-19 on this population will need to have a broad stakeholder engagement and address a wide range of health determinants. Peer-driven interventions have been effective for the prevention and control of infectious diseases such as HIV, STIs among Latino populations. Strengthening the links between community members and these organizations and promoting inter-organizational coordination to meet syndemic health, behavioral, economic, and legal needs of Latino communities are essential elements to mitigate the impact of COVID-19 on this low-resource population. In direct response to the NOT-MD-20-022/PAR PA-18-935, our ongoing community-academic partnership proposes to evaluate "CRISOL Contigo," a multi-level intervention to address the needs created or magnified by the COVID-19 pandemic among Latino communities in Philadelphia. CRISOL Contigo includes a peer-driven program and mobilization of Latino-serving organizations. In aim 1, the investigative team will adapt an ongoing Popular Opinion Leader (POL) program to address the unique health, social, and economic needs related to COVID-19 and the SAVAME syndemic. In aim 2, the investigative team will assess the efficacy of CRISOL Contigo to improve COVID-19 related preventive health behaviors and use and access to COVID-19 related testing and care (co-primary outcomes). In aim 3, the investigative team will examine the impact of CRISOL Contigo on community assets, interagency collaborations, and coordination among the Latino-serving organizations in Philadelphia. There are almost 20 million Latino immigrants in the US, and they play a central role in sustaining the vital parts of the US economy Tailored, multi-level interventions that consider the unique needs of Latinos are urgently needed to mitigate the impact of this and future outbreaks of COVID-19 on this disadvantaged population.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Latino or Hispanic
* Living in Philadelphia

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University Dornsife School of Public Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Popular Opinion Leader (POL): After successful completion of the new COVID-19 training module, POLs will reach out to members of their social networks to model and diffuse social norms to reduce the risk of COVID-19 infection and transmission, screen for symptoms and counsel regarding COVID-19, SAVAME syndemic factors, and refer at-risk or affected individuals to appropriate community services (e.g. free COVID-19 testing and treatment, mental health services, substance use services, violence prevention, support groups, etc.).
  The first 300 community contacts will be invited to complete a baseline and 3-month follow up surveys (via internet or phone).
Period: Overall Study
Arm/Group | Community Popular Opinion Leader (POL)
Started | 178
Completed | 139
Not Completed | 39

BASELINE CHARACTERISTICS:
Groups:
- Community Popular Opinion Leader (POL): A community popular opinion leader (POL) based intervention to promote measures to reduce COVID-19 risk, transmission, access to testing and treatment, reduction of the impact of COVID-19, and addressing the Substance Abuse, Violence, HIV/AIDS, and MEntal health (SAVAME) syndemic in the community. POLs will interact within their networks counseling regarding COVID-19 and SAVAME factors. The POLs will refer individuals to appropriate community services. POLs will record basic sociodemographic characteristics of all community contacts, the issue addressed, and their response to it. The first 300 community contacts will be invited to complete a baseline and 3-month follow up surveys (via internet or phone). The content of the surveys includes: 1) COVID-19 related questions (knowledge, impact, symptoms, risk factors, access to testing and care, acceptability contact tracing, vaccine) 2) Biological risk factors, 3) Social determinants of health, 4) SAVAME outcomes and access to services.
Arm/Group | Community Popular Opinion Leader (POL)
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino Black | 4
  Latino White | 12
  Latino Other | 119
  Latino Native American | 11
  Prefer not to answer, Unknown, More than one | 39
Region of Enrollment [Number; unit: participants]
  United States | 178
Education Category [Count of Participants; unit: Participants]
  Primary or below | 33
  More than Primary & <= High School | 111
  High school or more | 32
  Missing | 2
Baseline Income Category [Count of Participants; unit: Participants] — Self reported total monthly household income of all family members from all sources after taxes
  Participants
    <$1000 usd | 86
    $1000-$2000 usd | 38
    >$2000 usd | 21
    Missing/Don't know | 33
Prevalence of COVID-19 positive [Count of Participants; unit: Participants] — Defined as ever having a COVID-19 positive, doctor diagnosis or belief.
  Participants | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Five Protective COVID-19 Risk Measures
Description: This measure is the sum of the five protective COVID-19 risk measures: Use of mask, frequent hand washing, social distancing (including the ability to telework, and avoid crowded indoor spaces), and avoidance of contact with high-risk individuals. Scale ranged (0-5). The higher the score, the higher the number of protective behaviors
Time Frame: Baseline and 3 months
Population: Each of the rows indicates the mean (SD) of protective behaviors at baseline and 3 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Popular Opinion Leader (POL)
Number analyzed (Participants) | 139
score on a scale
  Baseline | 2.79 (1.23)
  3 Months | 2.66 (1.33)
Statistical Analysis 1: Comparison: Community Popular Opinion Leader (POL); This is a single-group study. Selected outcomes were measured at baseline (first interaction with the community popular opinion leader (POL) and 3 months after; Test type: Non-Inferiority — This is a single-group, of outcome measured at baseline and at 3 months. We hypothesized there would be an improvement or sustainability of the protective behaviours; p = 0.28, t-test, 2 sided; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.12 to 0.39], Standard Error of Mean 0.13

2. Primary Outcome: Number of Participants Who Lack Access to Health Care
Description: This measure is a composite dichotomous outcome variable, that indicates not having health insurance or not having a regular primary care provider.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Popular Opinion Leader (POL)
Number analyzed (Participants) | 139
Participants
  Baseline | 121
  3 Months | 122
Statistical Analysis 1: Comparison: Community Popular Opinion Leader (POL); Two sample test of proportions, testing whether the proportion of participants who lack health access at baseline and 3 months is equal (null hypothesis); Test type: Other — Test of proportions; p = 0.85, Test of proportions; difference in proportion = -0.007, 95% CI 2-sided [-0.08 to 0.07], Standard Error of Mean 0.04

3. Secondary Outcome: Number of Participants With SAVAME (Substance Abuse, Violence, HIV/AIDS, Mental Health)-Related Factors
Description: Substance abuse (yes/no), defined as binge drinking (>=4 or >=5 drinks on one occasion for women, and men, respectively), or use of drugs other than those required for medical reasons (at least once a week). Intimate partner violence (yes/no), defined as experiencing verbal or physical violence, categorized using answers to the following questions: In the 30 days, how often has a partner or spouse, "Yelled at you or said things to you that made you feel bad about yourself, embarrassed you in front of others, or frightened you?", "Done things like push, grab, hit, slap, kick, or throw things at you during an argument or because they were angry with you?". Any answer other than never was considered yes. HIV/AIDS (yes/no), defined as having a history of a positive test. Mental health (Yes/no), defined as depressive (CES-D-10 >=10) or anxiety (GAD-7 >=5) symptoms.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Popular Opinion Leader (POL)
Number analyzed (Participants) | 139
Participants
  Baseline | 64
  3 Months | 48
Statistical Analysis 1: Comparison: Community Popular Opinion Leader (POL); Test of proportions. Testing whether the proportion of participants who had a SAVAME factor at baseline and 3 months is equal (null hypothesis); Test type: Other — Test of proportions; p = 0.19, Test of proportions; difference in proportion = 0.07, 95% CI 2-sided [-0.04 to 0.19], Standard Error of Mean 0.58

4. Secondary Outcome: Lack of Access to SAVAME Services
Description: Self-report lack of access to any SAVAME (Substance abuse, Intimate partner violence, HIV/AIDS, or Mental health symptomatology) services, overall among all the participants
Time Frame: Baseline and 3 months
Population: Defined as self-report lack of access to any SAVAME services, overall among all the participants
Measure: Count of Participants; unit: Participants
Arm/Group | Community Popular Opinion Leader (POL)
Number analyzed (Participants) | 139
Participants
  Baseline | 52
  3 Months | 43
Statistical Analysis 1: Comparison: Community Popular Opinion Leader (POL); Test of proportions. Testing whether the proportion of participants who lack access to SAVAME related services at baseline and 3 months is equal (null hypothesis); Test type: Other — Test of proportions; p = 0.23, Test of proportions; difference in proportion = 0.067, 95% CI 2-sided [-0.04 to 0.18], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Community Popular Opinion Leader (POL)
All-Cause Mortality (participants affected / at risk) | 0/178
Serious Adverse Events (participants affected / at risk) | 0/178
Other Adverse Events (participants affected / at risk) | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT04646616/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT04646616/SAP_001.pdf